CLINICAL TRIAL: NCT00686374
Title: A Multi-center, Open-label Study of the Human Anti-TNF Monoclonal Antibody Adalimumab to Evaluate the Efficacy and the Long-term Safety and Tolerability of Repeated Administration of Adalimumab in Pediatric Subjects With Crohn's Disease Who Have Demonstrated a Clinical Response in the M06-806 Study
Brief Title: Efficacy and Long Term Safety of Adalimumab in Pediatric Subjects Who Have Demonstrated Clinical Response in M06-806
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M06-807; 2007-006494-90 (EudraCT Number)
Record Dates: First submitted 2008-05-27; First posted 2008-05-29 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; adalimumab
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Any adalimumab (Experimental): Adalimumab was administered via subcutaneous injection. Dosage was based on body weight and clinical status, and ranged from 10, 20, or 40 mg every other week to 20 or 40 mg every week.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Participants who enrolled into the study from blinded therapy in Study M06-806 received open-label (OL) therapy at a dose dependent on their body weight. Participants weighing ≥ 40 kg received 40 mg of adalimumab every other week (eow), and those who weighed < 40 kg received 20 mg of adalimumab eow. Starting at Week 8, participants who had a disease flare may have been switched to every week (ew) treatment at the same dose of adalimumab received while on eow treatment. Participants who enrolled from OL therapy in Study M06-806 continued to receive the same dose they were receiving (i.e., 40 mg ew or 20 mg ew) at the Week 52 visit of Study M06-806. Adalimumab dose could have been decreased to the next lower treatment level for those with body weight changes. Participants who responded to treatment may have also had their dosage frequency decreased from ew to eow dosing, as well as a decrease in dosage.
  Other Names: ABT-D2E7; Humira

SUMMARY:
This was a multicenter, open-label study to evaluate the human monoclonal anti-TNF-α antibody adalimumab as an effective therapy for maintaining clinical response in pediatric participants with Crohn's disease (CD) and to gather long-term safety and tolerability data in this population. Participants were allowed to enroll in the study if they participated in and successfully completed Study M06-806 (NCT00409682) through Week 52.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have successfully enrolled in and completed Study M06-806 through Week 52.
* Participant must have been a responder at any time point during the M06-806 study (defined as having achieved at least a 15-point reduction in the Pediatric Crohn's Disease Activity Index (PCDAI) from Baseline).
* If female, participants who were sexually active and of child-bearing potential were to be practicing an approved method of birth control throughout the study and for 150 days after study drug administration. Examples of approved methods of birth control included the following:

  1. Condoms, sponge, foam, jellies, diaphragm or intrauterine device (IUD)
  2. Oral, parenteral or intravaginal contraceptives
  3. A vasectomized partner
* Participant of legal age, parent or legal guardian, as required, voluntarily signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved informed consent form, after the nature of the study was explained and the participant of legal age, participant's parent, or legal guardian, as required, had the opportunity to ask questions. Participants were to be included in all discussions, and if required, their signature on an assent form was to be obtained.
* Parent or legal guardian of participant who was not of legal age, as required, must have been willing to actively supervise storage and administration of study drug and to ensure that the time of each dose was accurately recorded in the participant's diary.
* Participants of legal age, must have been willing to actively store, administer, and accurately record study drug administration in the participant diary.
* Participant was judged to be in acceptable medical condition, as determined by the Principal Investigator based upon results of clinical and laboratory evaluations done throughout the preceding Crohn's disease study M06-806.

Exclusion Criteria:

* For any reason, the participant was considered by the Investigator to be an unsuitable candidate for continuing therapy in the M06-807 study.
* Participant had abnormal laboratory or other test results that in the opinion of the Investigator would make the participant unsuitable to participate in this study.
* History of cancer or lymphoproliferative disease other than a successfully and completely treated cutaneous squamous cell or basal cell carcinoma or carcinoma in-situ of the cervix.
* History of listeriosis, histoplasmosis, chronic or active hepatitis B infection, human immunodeficiency virus (HIV) infection, any immunodeficiency syndrome, central nervous system (CNS) demyelinating disease or active TB (receiving treatment or not receiving treatment). Ongoing severe infections such as sepsis and opportunistic infections were exclusionary.
* Participant with known, symptomatic obstructive strictures.
* Participant who was planning surgical bowel resection at any time point while enrolled in the study.
* Participant who had short bowel syndrome as determined by the Investigator.
* Participant who was receiving total parenteral nutrition (TPN).
* Participant who was unwilling to discontinue growth hormone prior to the first dose of open-label study drug at the Baseline visit of M06-807.
* Female participant who was pregnant or currently breastfeeding.
* Participant with a history of clinically significant drug or alcohol abuse in the last year.
* Participant with a poorly controlled medical condition such as: uncontrolled diabetes, recurrent infections, unstable ischemic heart disease, moderate to severe heart failure, recent cerebrovascular accidents or any other condition which, in the opinion of the Investigator or the Sponsor, would put the participant at risk by participation in the protocol.
* Participant with any prior exposure to Tysabri (natalizumab).
* Participant with a known hypersensitivity to the excipients of adalimumab as stated in the label.
* Participant with a previous history of dysplasia of the gastrointestinal tract.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2008-05-01; Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Lazar, Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Faubion WA, Dubinsky M, Ruemmele FM, Escher J, Rosh J, Hyams JS, Eichner S, Li Y, Reilly N, Thakkar RB, Robinson AM, Lazar A. Long-term Efficacy and Safety of Adalimumab in Pediatric Patients with Crohn's Disease. Inflamm Bowel Dis. 2017 Mar;23(3):453-460. doi: 10.1097/MIB.0000000000001021. PMID 28129288
- [Derived] Horneff G, Seyger MMB, Arikan D, Kalabic J, Anderson JK, Lazar A, Williams DA, Wang C, Tarzynski-Potempa R, Hyams JS. Safety of Adalimumab in Pediatric Patients with Polyarticular Juvenile Idiopathic Arthritis, Enthesitis-Related Arthritis, Psoriasis, and Crohn's Disease. J Pediatr. 2018 Oct;201:166-175.e3. doi: 10.1016/j.jpeds.2018.05.042. Epub 2018 Jul 25. PMID 30054164
- [Derived] Ruemmele FM, Rosh J, Faubion WA, Dubinsky MC, Turner D, Lazar A, Eichner S, Maa JF, Alperovich G, Robinson AM, Hyams JS. Efficacy of Adalimumab for Treatment of Perianal Fistula in Children with Moderately to Severely Active Crohn's Disease: Results from IMAgINE 1 and IMAgINE 2. J Crohns Colitis. 2018 Nov 9;12(10):1249-1254. doi: 10.1093/ecco-jcc/jjy087. PMID 29939254
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 participants discontinued study drug when adalimumab became commercially available (received regulatory approval for pediatric Crohn's disease) in their country. These participants were considered to have completed the study, and are included as study completers in the subject disposition.
Period: Overall Study
Arm/Group | Any Adalimumab
Started | 100
Completed | 39
Not Completed | 61
Not completed — Lack of Efficacy | 10
Not completed — Adverse Event | 8
Not completed — Withdrew consent | 5
Not completed — Lost to Follow-up | 1
Not completed — Missing reason | 33
Not completed — Other, not specified | 4

BASELINE CHARACTERISTICS:
Population: ITT Population: all participants who received ≥ 1 dose of adalimumab in Study M06-807 and also had ≥ 1 non-missing efficacy measurement during the study.
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Study M06-806 Baseline
  years | 13.5 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 93
  Black | 3
  Other | 2
  Multi-race | 2
Body weight at Study M06-806 Baseline [Count of Participants; unit: Participants]
  < 40 kg | 38
  ≥ 40 kg | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Pediatric Crohn's Disease Activity Index (PCDAI) Clinical Remission Over Time
Description: Pediatric Crohn's Disease Activity Index (PCDAI) is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. Clinical remission was defined as PCDAI ≤ 10.
Time Frame: Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 100
Participants
  Week 0 | 67
  Week 4: number analyzed (Participants) | 98
  Week 4 | 65
  Week 8: number analyzed (Participants) | 97
  Week 8 | 67
  Week 12: number analyzed (Participants) | 96
  Week 12 | 60
  Week 24: number analyzed (Participants) | 94
  Week 24 | 59
  Week 36: number analyzed (Participants) | 87
  Week 36 | 60
  Week 48: number analyzed (Participants) | 82
  Week 48 | 54
  Week 60: number analyzed (Participants) | 79
  Week 60 | 60
  Week 72: number analyzed (Participants) | 76
  Week 72 | 49
  Week 84: number analyzed (Participants) | 74
  Week 84 | 54
  Week 96: number analyzed (Participants) | 77
  Week 96 | 54
  Week 108: number analyzed (Participants) | 72
  Week 108 | 54
  Week 120: number analyzed (Participants) | 67
  Week 120 | 52
  Week 144: number analyzed (Participants) | 64
  Week 144 | 51
  Week 168: number analyzed (Participants) | 58
  Week 168 | 44
  Week 192: number analyzed (Participants) | 55
  Week 192 | 44
  Week 216: number analyzed (Participants) | 50
  Week 216 | 36
  Week 240: number analyzed (Participants) | 46
  Week 240 | 37
  Week 264: number analyzed (Participants) | 37
  Week 264 | 31
  Week 288: number analyzed (Participants) | 29
  Week 288 | 24
  Week 312: number analyzed (Participants) | 18
  Week 312 | 14
  Week 336: number analyzed (Participants) | 11
  Week 336 | 8
  Week 360: number analyzed (Participants) | 8
  Week 360 | 7
  Week 384: number analyzed (Participants) | 2
  Week 384 | 2
  Week 408: number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Clinical Response as Defined by Pediatric Crohn's Disease Activity Index (PCDAI) Score Over Time
Description: Pediatric Crohn's Disease Activity Index (PCDAI) is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. The baseline PCDAI value was defined as the last non-missing value on or before the date of the first dose of study drug during Study M06-806. Clinical response was defined as a PCDAI ≥ 15 points lower than the Study M06-806 baseline PCDAI value.
Time Frame: Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 100
Participants
  Week 0 | 95
  Week 4: number analyzed (Participants) | 98
  Week 4 | 90
  Week 8: number analyzed (Participants) | 97
  Week 8 | 92
  Week 12: number analyzed (Participants) | 96
  Week 12 | 87
  Week 24: number analyzed (Participants) | 94
  Week 24 | 88
  Week 36: number analyzed (Participants) | 87
  Week 36 | 82
  Week 48: number analyzed (Participants) | 82
  Week 48 | 74
  Week 60: number analyzed (Participants) | 79
  Week 60 | 76
  Week 72: number analyzed (Participants) | 76
  Week 72 | 72
  Week 84: number analyzed (Participants) | 74
  Week 84 | 69
  Week 96: number analyzed (Participants) | 77
  Week 96 | 72
  Week 108: number analyzed (Participants) | 72
  Week 108 | 70
  Week 120: number analyzed (Participants) | 67
  Week 120 | 65
  Week 144: number analyzed (Participants) | 64
  Week 144 | 64
  Week 168: number analyzed (Participants) | 58
  Week 168 | 53
  Week 192: number analyzed (Participants) | 55
  Week 192 | 52
  Week 216: number analyzed (Participants) | 50
  Week 216 | 46
  Week 240: number analyzed (Participants) | 46
  Week 240 | 43
  Week 264: number analyzed (Participants) | 37
  Week 264 | 35
  Week 288: number analyzed (Participants) | 29
  Week 288 | 28
  Week 312: number analyzed (Participants) | 18
  Week 312 | 15
  Week 336: number analyzed (Participants) | 11
  Week 336 | 10
  Week 360: number analyzed (Participants) | 8
  Week 360 | 8
  Week 384: number analyzed (Participants) | 2
  Week 384 | 2
  Week 408: number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants Who Were in Crohn's Disease Activity Index (CDAI) Clinical Remission Over Time
Description: The CDAI includes 8 variables encompassing both subject-reported (symptoms, general well-being) and objective (medication usage, laboratory variables, presence of abdominal mass or complications, and weight) variables. For symptoms scores, participants kept track of daily symptoms on a diary card, and the daily symptom scores were summed for the week. Each item in the CDAI is assigned a specific weight, and the weighted values of the items are totaled to produce the CDAI score. Higher CDAI scores indicate greater disease activity; 0 is the lower limit with no set upper limit. The scale for the score is as follows: < 150 to indicate remission, 150 - 219 to define mildly active disease, 220 - 450 to define moderately active disease, and > 450 to define severely active disease. A CDAI was calculated at each visit for participants who were age 13 or older at Study M06-806 entry. The Study M06-806 Week 52 visit served as the baseline visit for this study.
Time Frame: Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408
Population: Participants ≥ 13 years old at Study M06-806 entry who received ≥ 1 dose of adalimumab in Study M06-807 and also had ≥ 1 non-missing efficacy measurement during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 65
Participants
  Week 0 | 58
  Week 4: number analyzed (Participants) | 63
  Week 4 | 55
  Week 8: number analyzed (Participants) | 62
  Week 8 | 58
  Week 12: number analyzed (Participants) | 61
  Week 12 | 53
  Week 24: number analyzed (Participants) | 59
  Week 24 | 54
  Week 36: number analyzed (Participants) | 55
  Week 36 | 52
  Week 48: number analyzed (Participants) | 53
  Week 48 | 48
  Week 60: number analyzed (Participants) | 52
  Week 60 | 49
  Week 72: number analyzed (Participants) | 50
  Week 72 | 47
  Week 84: number analyzed (Participants) | 50
  Week 84 | 46
  Week 96: number analyzed (Participants) | 50
  Week 96 | 45
  Week 108: number analyzed (Participants) | 49
  Week 108 | 45
  Week 120: number analyzed (Participants) | 43
  Week 120 | 42
  Week 144: number analyzed (Participants) | 41
  Week 144 | 40
  Week 168: number analyzed (Participants) | 35
  Week 168 | 35
  Week 192: number analyzed (Participants) | 33
  Week 192 | 31
  Week 216: number analyzed (Participants) | 30
  Week 216 | 27
  Week 240: number analyzed (Participants) | 29
  Week 240 | 26
  Week 264: number analyzed (Participants) | 24
  Week 264 | 23
  Week 288: number analyzed (Participants) | 18
  Week 288 | 17
  Week 312: number analyzed (Participants) | 15
  Week 312 | 15
  Week 336: number analyzed (Participants) | 9
  Week 336 | 8
  Week 360: number analyzed (Participants) | 7
  Week 360 | 7
  Week 384: number analyzed (Participants) | 1
  Week 384 | 1
  Week 408: number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants Who Were in Crohn's Disease Activity Index (CDAI) Clinical Response Over Time
Description: The CDAI includes 8 variables: subject-reported (symptoms, general well-being) and objective (medication usage, laboratory variables, presence of abdominal mass or complications, and weight). Participants kept track of symptoms on a diary card, and scores were summed for the week. Each item is assigned a specific weight, and the weighted values of the items are totaled to produce the CDAI score. Higher CDAI scores indicate greater disease activity; 0 is the lower limit with no set upper limit. Scale: < 150 (remission), 150 - 219 (mildly active disease), 220 - 450 (moderately active disease), and > 450 (severely active disease). A CDAI was calculated at each visit for participants ≥ 13 yrs old at M06-806 entry. Clinical response was defined as a decrease from M06-806 Baseline CDAI value of ≥ 70 pts. The M06-806 Baseline value was defined as the last non-missing value on or before the date of the 1st dose of study drug in M06-806.
Time Frame: Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384, 408
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 64
Participants
  Week 0 | 55
  Week 4: number analyzed (Participants) | 63
  Week 4 | 56
  Week 8: number analyzed (Participants) | 62
  Week 8 | 56
  Week 12: number analyzed (Participants) | 61
  Week 12 | 51
  Week 24: number analyzed (Participants) | 59
  Week 24 | 52
  Week 36: number analyzed (Participants) | 55
  Week 36 | 53
  Week 48: number analyzed (Participants) | 53
  Week 48 | 48
  Week 60: number analyzed (Participants) | 52
  Week 60 | 48
  Week 72: number analyzed (Participants) | 50
  Week 72 | 45
  Week 84: number analyzed (Participants) | 50
  Week 84 | 47
  Week 96: number analyzed (Participants) | 50
  Week 96 | 45
  Week 108: number analyzed (Participants) | 49
  Week 108 | 47
  Week 120: number analyzed (Participants) | 43
  Week 120 | 40
  Week 144: number analyzed (Participants) | 41
  Week 144 | 41
  Week 168: number analyzed (Participants) | 35
  Week 168 | 34
  Week 192: number analyzed (Participants) | 33
  Week 192 | 33
  Week 216: number analyzed (Participants) | 30
  Week 216 | 28
  Week 240: number analyzed (Participants) | 29
  Week 240 | 28
  Week 264: number analyzed (Participants) | 24
  Week 264 | 24
  Week 288: number analyzed (Participants) | 18
  Week 288 | 18
  Week 312: number analyzed (Participants) | 15
  Week 312 | 15
  Week 336: number analyzed (Participants) | 9
  Week 336 | 9
  Week 360: number analyzed (Participants) | 7
  Week 360 | 7
  Week 384: number analyzed (Participants) | 1
  Week 384 | 1
  Week 408: number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants in Steroid-free Pediatric Crohn's Disease Activity Index (PCDAI) Remission Over Time
Description: Pediatric Crohn's Disease Activity Index (PCDAI) is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. PCDAI corticosteroid-free remission was defined as discontinued corticosteroid use at least 90 consecutive days prior to the respective visit, with a PCDAI ≤ 10 at that visit.
Time Frame: Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384
Population: Participants with corticosteroid use at Study M06-806 entry who received ≥ 1 dose of adalimumab in Study M06-807 and also had ≥ 1 non-missing efficacy measurement during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 37
Participants
  Week 0 | 23
  Week 4 | 23
  Week 8 | 23
  Week 12 | 20
  Week 24 | 21
  Week 36: number analyzed (Participants) | 33
  Week 36 | 19
  Week 48: number analyzed (Participants) | 32
  Week 48 | 19
  Week 60: number analyzed (Participants) | 30
  Week 60 | 24
  Week 72: number analyzed (Participants) | 28
  Week 72 | 17
  Week 84: number analyzed (Participants) | 29
  Week 84 | 19
  Week 96: number analyzed (Participants) | 29
  Week 96 | 20
  Week 108: number analyzed (Participants) | 27
  Week 108 | 18
  Week 120: number analyzed (Participants) | 25
  Week 120 | 19
  Week 144: number analyzed (Participants) | 24
  Week 144 | 17
  Week 168: number analyzed (Participants) | 22
  Week 168 | 16
  Week 192: number analyzed (Participants) | 19
  Week 192 | 15
  Week 216: number analyzed (Participants) | 19
  Week 216 | 13
  Week 240: number analyzed (Participants) | 16
  Week 240 | 13
  Week 264: number analyzed (Participants) | 13
  Week 264 | 11
  Week 288: number analyzed (Participants) | 10
  Week 288 | 9
  Week 312: number analyzed (Participants) | 5
  Week 312 | 5
  Week 336: number analyzed (Participants) | 3
  Week 336 | 2
  Week 360: number analyzed (Participants) | 2
  Week 360 | 1
  Week 384: number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants in Steroid-free Crohn's Disease Activity Index (CDAI) Remission Over Time
Description: The CDAI includes 8 variables encompassing subject-reported (symptoms, general well-being) and objective (medication usage, laboratory variables, presence of abdominal mass or complications, and weight) variables. Participants kept track of daily symptoms on a diary card, and the scores were summed for the week. Each item in the CDAI is assigned a specific weight, and the items are totaled to produce the CDAI score. Higher CDAI scores indicate greater disease activity; 0 is the lower limit with no set upper limit. The scale for the score is as follows: < 150 (remission), 150 - 219 (mildly active disease), 220 - 450 (moderately active disease), and > 450 (severely active disease). A CDAI was calculated at each visit for subjects ≥ 13 years old at M06-806 entry. CDAI corticosteroid-free remission was defined as discontinued use at least 90 consecutive days prior to the respective visit and a CDAI < 150 at that visit.
Time Frame: Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384
Population: Participants ≥ 13 years old with corticosteroid use at Study M06-806 entry who received ≥ 1 dose of adalimumab in Study M06-807 and also had ≥ 1 non-missing efficacy measurement during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 26
Participants
  Week 0 | 21
  Week 4 | 22
  Week 8 | 22
  Week 12 | 20
  Week 24 | 21
  Week 36: number analyzed (Participants) | 24
  Week 36 | 22
  Week 48: number analyzed (Participants) | 24
  Week 48 | 22
  Week 60: number analyzed (Participants) | 23
  Week 60 | 21
  Week 72: number analyzed (Participants) | 21
  Week 72 | 19
  Week 84: number analyzed (Participants) | 22
  Week 84 | 20
  Week 96: number analyzed (Participants) | 22
  Week 96 | 20
  Week 108: number analyzed (Participants) | 21
  Week 108 | 18
  Week 120: number analyzed (Participants) | 18
  Week 120 | 16
  Week 144: number analyzed (Participants) | 17
  Week 144 | 15
  Week 168: number analyzed (Participants) | 14
  Week 168 | 13
  Week 192: number analyzed (Participants) | 12
  Week 192 | 11
  Week 216: number analyzed (Participants) | 13
  Week 216 | 10
  Week 240: number analyzed (Participants) | 11
  Week 240 | 10
  Week 264: number analyzed (Participants) | 8
  Week 264 | 8
  Week 288: number analyzed (Participants) | 6
  Week 288 | 6
  Week 312: number analyzed (Participants) | 4
  Week 312 | 4
  Week 336: number analyzed (Participants) | 3
  Week 336 | 2
  Week 360: number analyzed (Participants) | 2
  Week 360 | 1
  Week 384: number analyzed (Participants) | 0

7. Secondary Outcome: Mean Change From Baseline in Pediatric Crohn's Disease Activity Index (PCDAI) Over Time
Description: Pediatric Crohn's Disease Activity Index (PCDAI) is an index used to measure disease activity of pediatric patients with Crohn's disease assessing abdominal pain, stool frequency, patient functioning, hematocrit, erythrocyte sedimentation rate, albumin, weight, height, abdomen, perirectal disease, and extraintestinal manifestations. It ranges from 0 to 100; higher scores indicate more active disease. The baseline value was defined as the last non-missing value on or before the date of the first dose of study drug in Study M06-806. Negative changes indicate reductions (improvement) in disease activity.
Time Frame: Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 100
units on a scale
  Week 0 | -29.95 (11.459)
  Week 4: number analyzed (Participants) | 98
  Week 4 | -30.15 (11.514)
  Week 8: number analyzed (Participants) | 97
  Week 8 | -30.7 (11.415)
  Week 12: number analyzed (Participants) | 96
  Week 12 | -29.19 (11.405)
  Week 24: number analyzed (Participants) | 94
  Week 24 | -29.84 (11.702)
  Week 36: number analyzed (Participants) | 87
  Week 36 | -30.89 (12.354)
  Week 48: number analyzed (Participants) | 82
  Week 48 | -30.73 (11.983)
  Week 60: number analyzed (Participants) | 79
  Week 60 | -32.78 (10.927)
  Week 72: number analyzed (Participants) | 76
  Week 72 | -31.15 (10.404)
  Week 84: number analyzed (Participants) | 74
  Week 84 | -32.94 (10.809)
  Week 96: number analyzed (Participants) | 77
  Week 96 | -31.14 (11.33)
  Week 108: number analyzed (Participants) | 72
  Week 108 | -33.54 (9.538)
  Week 120: number analyzed (Participants) | 67
  Week 120 | -33.36 (10.441)
  Week 144: number analyzed (Participants) | 64
  Week 144 | -34.38 (9.204)
  Week 168: number analyzed (Participants) | 58
  Week 168 | -32.57 (11.273)
  Week 192: number analyzed (Participants) | 55
  Week 192 | -33.00 (13.258)
  Week 216: number analyzed (Participants) | 50
  Week 216 | -31.95 (12.344)
  Week 240: number analyzed (Participants) | 46
  Week 240 | -34.18 (13.386)
  Week 264: number analyzed (Participants) | 37
  Week 264 | -35.00 (9.242)
  Week 288: number analyzed (Participants) | 29
  Week 288 | -35.95 (11.941)
  Week 312: number analyzed (Participants) | 18
  Week 312 | -33.19 (14.318)
  Week 336: number analyzed (Participants) | 11
  Week 336 | -35.23 (12.013)
  Week 360: number analyzed (Participants) | 8
  Week 360 | -38.75 (10.69)
  Week 384: number analyzed (Participants) | 2
  Week 384 | -46.25 (22.981)

8. Secondary Outcome: Mean Change From Baseline in Crohn's Disease Activity Index (CDAI) Over Time
Description: The CDAI includes 8 variables: participant-reported (symptoms, general well-being) and objective (medication usage, laboratory variables, presence of abdominal mass or complications, and weight) variables. Participants kept track of daily symptoms on a diary card, and the scores were summed for the week. Each item in the CDAI is assigned a specific weight, and the items are totaled to produce the CDAI score. Higher CDAI scores indicate greater disease activity; 0 is the lower limit with no set upper limit. The scale for the score is as follows: < 150 (remission), 150 - 219 (mildly active disease), 220 - 450 (moderately active disease) and > 450 (severely active disease). A CDAI was calculated at each visit for those who were ≥ 13 years old at Study M06-806 entry. The baseline value was defined as the last non-missing value on or before the date of the first dose of study drug in Study M06-806. Negative changes indicate reductions (improvement) in disease activity.
Time Frame: Week 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360, 384
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Any Adalimumab
Number analyzed (Participants) | 64
units on a scale
  Week 0 | -160.8 (82.543)
  Week 4: number analyzed (Participants) | 63
  Week 4 | -159.9 (79.986)
  Week 8: number analyzed (Participants) | 62
  Week 8 | -164.45 (79.272)
  Week 12: number analyzed (Participants) | 61
  Week 12 | -151.34 (87.157)
  Week 24: number analyzed (Participants) | 59
  Week 24 | -161.51 (84.663)
  Week 36: number analyzed (Participants) | 55
  Week 36 | -173.55 (77.358)
  Week 48: number analyzed (Participants) | 53
  Week 48 | -162.08 (86.292)
  Week 60: number analyzed (Participants) | 52
  Week 60 | -168.27 (82.605)
  Week 72: number analyzed (Participants) | 50
  Week 72 | -165.4 (80.038)
  Week 84: number analyzed (Participants) | 50
  Week 84 | -172.68 (86.223)
  Week 96: number analyzed (Participants) | 50
  Week 96 | -168.3 (79.658)
  Week 108: number analyzed (Participants) | 49
  Week 108 | -171.63 (85.19)
  Week 120: number analyzed (Participants) | 43
  Week 120 | -179.14 (86.93)
  Week 144: number analyzed (Participants) | 41
  Week 144 | -181.53 (78.99)
  Week 168: number analyzed (Participants) | 35
  Week 168 | -175.05 (80.965)
  Week 192: number analyzed (Participants) | 33
  Week 192 | -172.42 (76.381)
  Week 216: number analyzed (Participants) | 30
  Week 216 | -173.13 (78.588)
  Week 240: number analyzed (Participants) | 29
  Week 240 | -184.46 (94.114)
  Week 264: number analyzed (Participants) | 24
  Week 264 | -186.42 (75.396)
  Week 288: number analyzed (Participants) | 18
  Week 288 | -197.11 (88.029)
  Week 312: number analyzed (Participants) | 15
  Week 312 | -199.00 (77.184)
  Week 336: number analyzed (Participants) | 9
  Week 336 | -240.33 (97.395)
  Week 360: number analyzed (Participants) | 7
  Week 360 | -224.86 (89.025)
  Week 384: number analyzed (Participants) | 1
  Week 384 | -458.00

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration in Study M06-806 until 70 days after the last dose of study drug in Study M06-807 (up to 470 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) or serious adverse event (SAE) with an onset date that is after the first dose of study drug until 70 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Arm/Group | Any Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 48/100
Other Adverse Events (participants affected / at risk) | 98/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any Adalimumab (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 2
LYMPHADENITIS (Blood and lymphatic system disorders) | 1
VERTIGO (Ear and labyrinth disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 25
FAECAL VOLUME INCREASED (Gastrointestinal disorders) | 1
GASTRITIS (Gastrointestinal disorders) | 2
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1
ILEAL PERFORATION (Gastrointestinal disorders) | 1
ILEAL STENOSIS (Gastrointestinal disorders) | 1
LARGE INTESTINAL STENOSIS (Gastrointestinal disorders) | 1
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1
OESOPHAGITIS (Gastrointestinal disorders) | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1
SMALL INTESTINAL STENOSIS (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 1
FATIGUE (General disorders) | 1
PYREXIA (General disorders) | 1
HEPATITIS (Hepatobiliary disorders) | 1
ABDOMINAL ABSCESS (Infections and infestations) | 1
ANAL ABSCESS (Infections and infestations) | 3
CYSTITIS VIRAL (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 2
HERPES VIRUS INFECTION (Infections and infestations) | 1
IMPETIGO (Infections and infestations) | 1
PELVIC ABSCESS (Infections and infestations) | 1
PERIRECTAL ABSCESS (Infections and infestations) | 1
PERITONITIS (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 2
SALMONELLOSIS (Infections and infestations) | 1
SINUSITIS (Infections and infestations) | 1
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 1
SUBCUTANEOUS ABSCESS (Infections and infestations) | 2
TONSILLITIS (Infections and infestations) | 1
TOOTH ABSCESS (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
VIRAL INFECTION (Infections and infestations) | 1
YERSINIA INFECTION (Infections and infestations) | 1
BONE CONTUSION (Injury, poisoning and procedural complications) | 1
CONCUSSION (Injury, poisoning and procedural complications) | 1
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
HEART RATE IRREGULAR (Investigations) | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1
DIZZINESS (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
SCHIZOAFFECTIVE DISORDER (Psychiatric disorders) | 1
SOMATIC SYMPTOM DISORDER (Psychiatric disorders) | 1
SUICIDAL IDEATION (Psychiatric disorders) | 1
PELVIC FLUID COLLECTION (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any Adalimumab (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 8
LEUKOPENIA (Blood and lymphatic system disorders) | 5
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 7
PALPITATIONS (Cardiac disorders) | 5
EAR PAIN (Ear and labyrinth disorders) | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 24
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 15
ANAL FISSURE (Gastrointestinal disorders) | 9
CONSTIPATION (Gastrointestinal disorders) | 15
CROHN'S DISEASE (Gastrointestinal disorders) | 24
DIARRHOEA (Gastrointestinal disorders) | 26
DYSPEPSIA (Gastrointestinal disorders) | 5
HAEMATOCHEZIA (Gastrointestinal disorders) | 8
MALPOSITIONED TEETH (Gastrointestinal disorders) | 6
NAUSEA (Gastrointestinal disorders) | 19
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 5
TOOTHACHE (Gastrointestinal disorders) | 5
VOMITING (Gastrointestinal disorders) | 22
FATIGUE (General disorders) | 18
INJECTION SITE PAIN (General disorders) | 7
INJECTION SITE REACTION (General disorders) | 16
PAIN (General disorders) | 6
PYREXIA (General disorders) | 20
HYPERSENSITIVITY (Immune system disorders) | 5
SEASONAL ALLERGY (Immune system disorders) | 8
BRONCHITIS (Infections and infestations) | 11
CONJUNCTIVITIS (Infections and infestations) | 9
EAR INFECTION (Infections and infestations) | 10
EYE INFECTION (Infections and infestations) | 5
GASTROENTERITIS (Infections and infestations) | 7
GASTROENTERITIS VIRAL (Infections and infestations) | 7
HERPES ZOSTER (Infections and infestations) | 8
IMPETIGO (Infections and infestations) | 7
INFLUENZA (Infections and infestations) | 15
ORAL HERPES (Infections and infestations) | 5
OTITIS MEDIA (Infections and infestations) | 8
PHARYNGITIS (Infections and infestations) | 20
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 14
PNEUMONIA (Infections and infestations) | 8
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 5
RHINITIS (Infections and infestations) | 10
SINUSITIS (Infections and infestations) | 17
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 5
TONSILLITIS (Infections and infestations) | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 31
URINARY TRACT INFECTION (Infections and infestations) | 14
VIRAL INFECTION (Infections and infestations) | 18
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 39
CONTUSION (Injury, poisoning and procedural complications) | 6
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 9
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 6
ANTINUCLEAR ANTIBODY POSITIVE (Investigations) | 5
C-REACTIVE PROTEIN INCREASED (Investigations) | 15
RED BLOOD CELL SEDIMENTATION RATE INCREASED (Investigations) | 8
DECREASED APPETITE (Metabolism and nutrition disorders) | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 21
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 5
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 8
MYALGIA (Musculoskeletal and connective tissue disorders) | 9
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13
DIZZINESS (Nervous system disorders) | 6
HEADACHE (Nervous system disorders) | 37
MIGRAINE (Nervous system disorders) | 8
DEPRESSION (Psychiatric disorders) | 6
INSOMNIA (Psychiatric disorders) | 6
DYSMENORRHOEA (Reproductive system and breast disorders) | 7
COUGH (Respiratory, thoracic and mediastinal disorders) | 20
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 6
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 12
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 27
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 5
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 7
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 7
ACNE (Skin and subcutaneous tissue disorders) | 7
ALOPECIA (Skin and subcutaneous tissue disorders) | 5
DRY SKIN (Skin and subcutaneous tissue disorders) | 7
ECZEMA (Skin and subcutaneous tissue disorders) | 8
ERYTHEMA (Skin and subcutaneous tissue disorders) | 6
PSORIASIS (Skin and subcutaneous tissue disorders) | 5
RASH (Skin and subcutaneous tissue disorders) | 15
URTICARIA (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-05-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT00686374/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT00686374/SAP_001.pdf